CLINICAL TRIAL: NCT02434861
Title: An Open Label, Single Dose, Three Part Study to Assess the Effects of Rolapitant (1.8 mg/mL Rolapitant IV Solution) on the Pharmacokinetics of Digoxin (P-gp); Sulfasalazine (BCRP); and the Cooperstown Cocktail (Midazolam [CYP3A4], Omeprazole [CYP2C19], Warfarin [CYP2C9], Caffeine [CYP1A2], and Dextromethorphan [CYP2D6]) in Healthy Subjects
Brief Title: An Open Label, Single Dose, Three Part Study to Assess the Effects of Rolapitant (2 mg/mL IV Solution) on the Pharmacokinetics of Digoxin; Sulfasalazine; and the Cooperstown Cocktail (Midazolam, Omeprazole, Warfarin, Caffeine, and Dextromethorphan in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PR-11-5021-C
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — rolapitant; Digoxin; Sulfasalazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A (Experimental): Rolapitant IV and Digoxin
  Interventions: Drug: Rolapitant; Drug: Digoxin
- Part B (Experimental): Rolapitant IV and Sulfasalazine
  Interventions: Drug: Rolapitant; Drug: Sulfasalazine
- Part C (Experimental): Rolapitant IV and Cooperstown Cocktail
  Interventions: Drug: Rolapitant; Drug: Cooperstown Cocktail

INTERVENTIONS:
Drug: Rolapitant
Drug: Digoxin — P-gp substrate
  Arms: Part A
Drug: Sulfasalazine — BCRP substrate
  Arms: Part B
Drug: Cooperstown Cocktail — Midazolam, omeprazole, warfarin, caffeine, and dextromethorphan
  Arms: Part C

SUMMARY:
The objective of this Open Label Study is to evaluate effects of Rolapitant IV solution, and its metabolite, on the pharmacokinetics (PK) of the P-gp substrate (digoxin), the BCRP substrate (sulfasalazine), and multiple cytochrome P450 (CYP) probe substrates in a healthy adult population.

DETAILED DESCRIPTION:
* Part A will compare the PK of oral digoxin alone and in combination with an IV infusion of rolapitant.
* Part B will compare the PK of an oral dose of sulfasalazine alone to the PK of an oral dose of sulfasalazine in combination with an IV infusion of rolapitant
* Part C will compare the PK of an oral dose of the Cooperstown Cocktail (midazolam, omeprazole, warfarin, caffeine, and dextromethorphan) alone and when given in combination with an IV infusion of rolapitant.

ELIGIBILITY:
Main Inclusion Criteria:

* Subjects must be healthy males or females aged 18 to 55 years (inclusive)
* Female subjects (of childbearing potential) must have a negative pregnancy test at Screening and on Day -1
* Female subjects of childbearing potential must agree to use an accepted method of birth control (excluding hormonal birth control methods) before Visit 1 and to continue its use during the study and for at least 30 days after the final dose
* Subjects must have a body mass index (BMI) from 18.5 to 32.0 kg/m2 (inclusive) and a weight of ≥50 kg at Screening
* Subjects must be capable of understanding the informed consent after the risks and benefits of the study have been explained; subjects must be able to sign a written informed consent and be willing to comply with the protocol requirements
* Subjects must be in general good health as determined by the Investigator based on pre-study medical and surgical history, physical examination [PE], and clinical laboratory tests

Main Exclusion Criteria:

* Subjects who have participated in another investigational study within 30 days or 5 half-lives of the test drug's biologic activity, whichever is longer, before the time of the first study dose
* Subjects who have a history of relevant allergies (including asthma, food, or drug allergies) as determined by the Investigator
* Subjects who have had significant blood loss, or have donated or received ≥1 units (450 mL) of blood, within 30 days before the first study dose
* Subjects who have a history of hypersensitivity to rolapitant IV or any of its excipients or who have participated in a previous rolapitant study within 6 months prior to administration of the first dose of study drug (Day 1)
* Subjects with poor venous access and/or cannot tolerate venipuncture
* Subjects with a history of significant complications or anxiety associated with the IV administration of medications that, in the opinion of the Investigator, could make the subject
* Subjects who have a history of hypersensitivity to sulfasalazine (Part B only).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
AUC: area under the plasma concentration-time curve | Predose - up to 120 hours postdose
  To evaluate the effect of Rolapitant on the PK of probe substrates
Cmax = observed maximum plasma concentration | Predose - up to 120 hours postdose
  To evaluate the effect of Rolapitant on the PK of probe substrates

SECONDARY OUTCOMES:
Number of participants with adverse events | 0 - 38 days
  To evaluate the safety and tolerability of combination administration of the P-gp substrate (digoxin), the BCRP substrate (sulfasalazine), and CYP probe substrates (midazolam, omeprazole, warfarin, caffeine, and dextromethorphan [Cooperstown Cocktail]) with a single dose of rolapitant IV in a healthy adult population, as assessed by incidence and severity of AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Vargo, MD, Study Director — Tesaro, Inc.
Locations (1):
- Parexel Early Phase Unit, Baltimore, Maryland, United States